CLINICAL TRIAL: NCT04219787
Title: Swiss Multicenter Randomized Controlled Trial on Different Limb Lengths in Gastric Bypass Surgery
Brief Title: Different Limb Lengths in Gastric Bypass Surgery
Acronym: SLIM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clarunis - Universitäres Bauchzentrum Basel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-02392
Record Dates: First submitted 2020-01-03; First posted 2020-01-07 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Obesity, Morbid; Diabetes Mellitus, Type 2; Hypertension; Dyslipidemias; Sleep Apnea
Keywords: Roux-en-Y Gastric Bypass; Biliopancreatic Limb Length
MeSH Terms: conditions — Obesity, Morbid; Diabetes Mellitus, Type 2; Hypertension; Dyslipidemias; Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long Biliopancreatic Limb LRYGB (Experimental): LRYGB with an 180 cm biliopancreatic limb (BPL) and an alimentary limb (AL) of 80 cm.
  Interventions: Procedure: Long BPL LRYGB
- Short Biliopancreatic Limb LRYGB (Active Comparator): Standard LRYGB with a 80 cm BPL and a 180 cm long AL.
  Interventions: Procedure: Short BPL LRYGB

INTERVENTIONS:
Procedure: Long BPL LRYGB — LRYGB with an 180 cm BPL and an AL of 80 cm.
  Other Names: LBPL LRYGB
  Arms: Long Biliopancreatic Limb LRYGB
Procedure: Short BPL LRYGB — The second group will receive a standard LRYGB with a 80 cm BPL and a 180 cm long AL.
  Other Names: SBPL LRYGB
  Arms: Short Biliopancreatic Limb LRYGB

SUMMARY:
Obesity and type 2 diabetes mellitus (T2DM) are reaching epidemic proportions in the developed world. In morbidly obese patients only surgical treatment (bariatric operations) leads to a sustained weight loss and relief of co-morbidities in the majority of patients. One of the most frequently performed operations is the laparoscopic proximal Roux-en-Y gastric bypass (LRYGB). There is still lack of knowledge why some patients respond much better than others to an identically performed procedure. Therefore, a number of variations of this operation have been introduced over the past 50 years. Increasing the length of small bowel being bypassed has the potential to improve the effect of the operation but buries the risk of nutrient deficiencies. The metabolic effect of LRYGB occurs, in part, independently of weight loss. The mechanisms underlying metabolic improvement through metabolic surgery are not yet fully understood.

ELIGIBILITY:
Inclusion Criteria:

* informed consent as documented by signature
* patients with BMI of 35 kg/m2 or higher who comply with the regulatory rules for bariatric surgery in Switzerland

Exclusion Criteria:

* general contraindications to kind of surgery
* known or suspected non-compliance, drug or alcohol abuse
* inability to follow the procedures of the study, e.g. due to language problems, psychological disorders etc. of the participant
* participation in another study
* age < 18 years or > 65 years
* BMI > 60 kg/m2
* height < 145 cm
* CL length of < 180 cm as measured intraoperatively
* ASA physical status classification > III
* inflammatory bowel disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint | From baseline to 5 years after surgery.
  Percent total weight loss (%TWL, superiority), while not leading to a larger nutritional de- ficiency rate (non-inferiority).

SECONDARY OUTCOMES:
Secondary endpoints | From baseline to 5 years after surgery.
  Percent excess body mass index loss (%EBMIL), remission of comorbidities, complication rate/safety, and quality of life 1, 3, and 5 years after long and short BPL RYGB.

CONTACTS AND LOCATIONS:
Overall Officials: Marko Kraljevic, MD, Study Chair — Clarunis - Universitäres Bauchzentrum Basel; Marco Bueter, MD, Professor, Study Chair — University Hospital Zurch
Locations (1):
- Clarunis University Center for Gastrointestinal and Liver Diseases, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kraljevic M, Schneider R, Wolnerhanssen B, Bueter M, Delko T, Peterli R. Different limb lengths in gastric bypass surgery: study protocol for a Swiss multicenter randomized controlled trial (SLIM). Trials. 2021 May 19;22(1):352. doi: 10.1186/s13063-021-05313-6. PMID 34011386